CLINICAL TRIAL: NCT03195946
Title: Interventional, Open-label, Multiple-dose Study to Investigate the Effects of Multiple Doses of Lu AF35700 on the Pharmacokinetics of Cytochrome P450 (CYP450) Substrates Dextromethorphan (CYP2D6), Caffeine (CYP1A2), Omeprazole (CYP2C19), and Midazolam (CYP3A4/5) in Healthy Young Adults
Brief Title: Effects of Repeated Doses of Lu AF35700 on Drug Metabolizing Enzymes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200A; 2016-003187-39 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Lu AF35700; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF35700 and Cocktail of CYP450 substrates (Experimental): Day 1 oral midazolam administration, Day 2 Cocktail of CYP450 substrates administration. Daily Lu AF35700 administration from Day 5 to Day 28 with co-administration on Day 27 with oral midazolam and Day 28 with CYP450 substrate cocktail
  Interventions: Drug: Lu AF35700; Drug: Midazolam; Drug: Cocktail of CYP450 substrates

INTERVENTIONS:
Drug: Lu AF35700 — tablets for oral use, 10 mg/day
Drug: Midazolam — syrup for oral use, 4mg/day
Drug: Cocktail of CYP450 substrates — Caffeine tablets for oral use, 200 mg/day. Omeprazole tablets for oral use, 40 mg/day. Dextromethorphan tablets for oral use, 30 mg/day. Midazolam IV solution for Intravenous use, 0.025 mg/kg/day

SUMMARY:
This study will help determine which types of drugs that may interact with Lu AF35700

ELIGIBILITY:
Inclusion Criteria:

* Body weight at least 50 kg and Body Mass Index 19 - 30 kg/m2
* Good general health ascertained by a detailed medical history, laboratory tests and physical examination

Exclusion Criteria:

-Pregnant or lactating women

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf): Area under the plasma concentration-time curve from zero to infinity | Up to 24 hours post dose on the following days: Day 1 and 27 for oral midazolam. Day 2 and 28 for cocktail components.
  Area under the plasma concentration-time curve from zero to infinity for oral midazolam and metabolite and all drug cocktail components and their metabolites
Cmax: Maximum observed concentration | Up to 24 hours post dose on the following days: Day 1 and 27 for oral midazolam. Day 2 and 28 for Cocktail components.
  Maximum observed concentration of oral midazolam and all drug cocktail components and their metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No